CLINICAL TRIAL: NCT02421328
Title: Comparative Study of the Effects of Continuous Positive Airway Pressure and Heated, Humidified High Flow Nasal Cannula on Diaphragmatic Dimensions in Preterm Infants
Brief Title: Study of the Effects of CPAP and HHHFNC on Diaphragmatic Dimensions in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University Children Hospital (Other)
Responsible Party: Principal Investigator, Hesham Abdel-Hady, Professor of Pediatrics, Mansoura University Children Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MS 874
Record Dates: First submitted 2015-04-13; First posted 2015-04-20 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Respirtory Distress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CPAP first (Active Comparator): Infant will be given nasal CPAP for 60 minutes and then put on HHHFNC for another 60 minutes. Ultrasonographic assessment of diaphragmatic dimensions and excursion will be done at the end of the 60 minute periods on nasal CPAP and HHHFNC. After the 2 h study period (2×60 minutes epochs) further respiratory support will be at the discretion of the clinical team
  Interventions: Device: CPAP first (Fisher & Paykel Healthcare)
- HHHFNC first (Active Comparator): Infant will be given HHHFNC for 60 minutes and then switched to nasal CPAP for another 30 minutes. Ultrasonographic assessment of diaphragmatic dimensions and excursion will be done at the end of the 60 minute periods on HHHFNC and nasal CPAP. After the 2 h study period (2×60 minutes epochs) further respiratory support will be at the discretion of the clinical team
  Interventions: Device: HHHFNC first (Fisher & Paykel Healthcare)

INTERVENTIONS:
Device: CPAP first (Fisher & Paykel Healthcare) — Infants will start on nasal CPAP for 60 minutes and then switched to HHHFNC for anther 60 minutes. Ultrasonographic assessment of diaphragmatic dimensions and excursion will be done at the end of each 60 minute epochs.
  Arms: CPAP first
Device: HHHFNC first (Fisher & Paykel Healthcare) — Infants will start on HHHFNC for 60 minutes and then switched to nasal CPAP for anther 60 minutes. Ultrasonographic assessment of diaphragmatic dimensions and excursion will be done at the end of each 60 minute epochs.
  Arms: HHHFNC first

SUMMARY:
This is a prospective, randomized crossover study to recognize the effects of nasal continuous positive airway pressure (CPAP) versus heated humidified high flow nasal cannula (HHHFNC) on diaphragmatic dimensions and excursion (evaluated by ultrasonography) in preterm infants.

DETAILED DESCRIPTION:
Preterm infants will be recruited consecutively from NICU of Mansoura University Children's Hospital. They will be randomized in two groups; one group will start on nasal CPAP (Fisher & Paykel Healthcare, Auckland, New Z ealand) (Pressure 5 cmH2O) for 60 minutes and then will be switched to HHHFNC (Fisher & Paykel Healthcare, Auckland, New Z ealand) (flow of 4 l/m) for another 60 minutes. The other group will start on HHHFNC and then switched to nasal CPAP.

After the 2 h study period (2×60 minutes epochs) further respiratory support will be at the discretion of the clinical team.

Ultrasonographic assessment of diaphragmatic dimensions and excursion will be analyzed in different respiratory cycles and the average of 3 cycles will be calculated at the end of the 60 minutes periods on nasal CPAP and HHHFNC.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants < 37 weeks.
* Stable on nasal continuous positive airway pressure (CPAP) for at least 24 hours.
* On less than 35% oxygen.

Exclusion Criteria:

* Congenital and acquired problems of the gastrointestinal tract as necrotizing enterocolitis, esophageal perforation and tracheoesophageal fistula.
* Phrenic nerve injury and/or diaphragm paralysis
* Congenital/acquired neurological deficit and/or seizures
* Hemodynamic instability
* Congenital heart disease (including symptomatic patent ductus arteriosus)
* Undergoing treatment for sepsis or pneumonia.
* Use of muscle relaxants, narcotic analgesics, or gastric motility agents.
* Congenital anomalies of respiratory tract.
* Infants requiring more than 35% oxygen.
* Infants with facial anomalies.
* Infants with pneumothorax and/or pneumomediatinum.
* Infants in the immediate postoperative period.
* Infants with significant gastric residues and vomiting.

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic dimensions (inspiratory diaphragmatic thickness, expiratory diaphragmatic thickness and delta diaphragmatic thickness) | at the end of each 60 minutes epoch on nasal CPAP
  Ultrasonographic assessment of (inspiratory diaphragmatic thickness, expiratory diaphragmatic thickness and delta diaphragmatic thickness will be assessed at the end of each 60 minutes epoch on nasal CPAP. Diaphragm thickness will be measured as the perpendicular distance between the pleural and peritoneal reflections. All measurements will be performed during quiet breathing. Several respiratory cycles will be recorded, and measurements will be averaged from at least three different cycles.
Right and left diaphragmatic excursion | at the end of each 60 minute epoch on CPAP
  Ultrasonographic assessment of right and left diaphragmatic excursion will be assessed at the end of each 60 minutes epoch on nasal CPAP. The displacements of the liver and spleen will be monitored in real-time. Using M-mode ultrasonography, with the probe fixed on the chest wall during respiration, ultrasonographic image of will be frozen and a mark for measurement will be placed on the image at the location of the most caudal margin of the liver or spleen at the end of expiration, and a second mark will be placed on the new location of the most caudal margin of the liver or spleen at the end of inspiration. The distance between the two marks will be then measured and defined as the displacement of the liver or the spleen (right or left diaphragmatic excursion). Several respiratory cycles will be recorded, and measurements will be averaged from at least three different cycles.
Diaphragmatic dimensions (inspiratory diaphragmatic thickness, expiratory diaphragmatic thickness and delta diaphragmatic thickness) | at the end of each 60 minutes epochs on HHHNC
  Ultrasonographic assessment of (inspiratory diaphragmatic thickness, expiratory diaphragmatic thickness and delta diaphragmatic thickness will be assessed at the end of each 60 minutes epoch on HHHFNC. Diaphragm thickness will be measured as the perpendicular distance between the pleural and peritoneal reflections. All measurements will be performed during quiet breathing. Several respiratory cycles will be recorded, and measurements will be averaged from at least three different cycles.
Right and left diaphragmatic excursion | at the end of each 60 minutes epochs on HHHNC
  Ultrasonographic assessment of right and left diaphragmatic excursion will be assessed at the end of each 60 minutes epoch on HHHFNC. The displacements of the liver and spleen will be monitored in real-time. Using M-mode ultrasonography, with the probe fixed on the chest wall during respiration, ultrasonographic image of will be frozen and a mark for measurement will be placed on the image at the location of the most caudal margin of the liver or spleen at the end of expiration, and a second mark will be placed on the new location of the most caudal margin of the liver or spleen at the end of inspiration. The distance between the two marks will be then measured and defined as the displacement of the liver or the spleen (right or left diaphragmatic excursion). Several respiratory cycles will be recorded, and measurements will be averaged from at least three different cycles.

SECONDARY OUTCOMES:
Respiratory rate | At the end of each 60 minutes epochs on CPAP and HHHFNC
  Respiratory rate will be assessed at the end of each 60 minutes epoch on CPAP or HHHFNC
Heart rate | At the end of each 60 minutes epochs on CPAP and HHHFNC
  Heart rate will be assessed at the end of each 60 minutes epoch on CPAP or HHHFNC
Spo2 | At the end of each 60 minutes epochs on CPAP and HHHFNC
  Oxygen saturation by pulse oximetry (SpO2) will be assessed at the end of each 60 minutes epoch on CPAP or HHHFNC
Number of apneas | during the 60 minutes epochs on CPAP and HHHFNC
  Number of apneas will be recorded during the 60 minutes epoch on CPAP or HHHFNC

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Neonatal Intensive Care Unit, Mansoura University Children Hospital, Al Mansurah, Dakahlia Governorate
  - NICU, Mansoura University Children's Hospital, Al Mansurah, Dakahlia Governorate

REFERENCES:
- [Derived] El-Mogy M, El-Halaby H, Attia G, Abdel-Hady H. Comparative Study of the Effects of Continuous Positive Airway Pressure and Nasal High-Flow Therapy on Diaphragmatic Dimensions in Preterm Infants. Am J Perinatol. 2018 Apr;35(5):448-454. doi: 10.1055/s-0037-1608682. Epub 2017 Nov 13. PMID 29132179